CLINICAL TRIAL: NCT04641975
Title: A Phase 3, Double-blind, Randomized, Multicenter, Parallel Group, Placebo-controlled Sequential Dose Titration Study to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Pediatric Subjects From 5 to < 18 Years of Age With Overactive Bladder
Brief Title: A Study to Evaluate Mirabegron in Pediatric Participants From 5 to Less Than 18 Years of Age With Overactive Bladder (OAB)
Acronym: Dolphin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termination due to operational futility
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 178-CL-204; 2016-001767-37 (EudraCT Number)
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Results first posted 2023-12-28 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Overactive Bladder (OAB); Pharmacokinetics of Mirabegron
Keywords: Pediatrics; mirabegron
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Mirabegron (5 to <12 Years) (Experimental): Participants aged 5 to < 12 years received initial dose of 25 milligram (mg) of mirabegron orally once daily based on weight (pediatric equivalent dose of 25 mg [PED25]) on day 1. Participants with a body weight ≥ 35 kilogram (kg) received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the pediatric equivalent dose of 50 mg [PED50] based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
  Interventions: Drug: Mirabegron
- Placebo (5 to <12 Years) (Placebo Comparator): Participants aged 5 to < 12 years received placebo matched to mirabegron orally once daily based on weight PED25 on day 1. Participants with a body weight ≥ 35 kg received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the PED50 based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
  Interventions: Drug: Placebo
- Mirabegron (12 to <18 Years) (Experimental): Participants aged 12 to < 18 years received initial dose of 25 mg of mirabegron orally once daily based on weight PED25 on day 1. Participants with a body weight ≥ 35 kg received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the PED50 based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
  Interventions: Drug: Mirabegron
- Placebo (12 to <18 Years) (Placebo Comparator): Participants aged 12 to < 18 years received placebo matched to mirabegron orally once daily based on weight PED25 on day 1. Participants with a body weight ≥ 35 kg received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the PED50 based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron — Oral/ Oral Suspension: Participants with a body weight of ≥ 35 kg are to receive the tablet form of IP unless unable to swallow tablets and will be provided the oral suspension as an alternative. Participants with a body weight < 35 kg or those who cannot be dosed with the tablet will receive oral suspension.
  Other Names: Betanis; Betmiga; Myrbetriq; YM178
  Arms: Mirabegron (12 to <18 Years); Mirabegron (5 to <12 Years)
Drug: Placebo — Oral/ Oral Suspension
  Arms: Placebo (12 to <18 Years); Placebo (5 to <12 Years)

SUMMARY:
The purpose of this study was to evaluate the efficacy of mirabegron in children (5 to < 12 years of age) with OAB.

This study will also evaluated the safety and tolerability of mirabegron in pediatric participants with OAB and evaluated the pharmacokinetics after multiple dose administration of mirabegron in pediatric participants with OAB.

DETAILED DESCRIPTION:
The study consisted of 3 periods (Screening period/urotherapy (4 weeks); Double-blind, placebo-controlled period (12 weeks); Follow-up period (2 weeks)) for a total duration of 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has OAB defined according to the International Children's Continence Society (ICCS) criteria.
* Subject weighs at least 13 kg at screening.
* Subject is able to take the IP in accordance with the protocol.
* Subject agrees to drink an adequate fluid volume during urine collection weekends.
* Subject and subject's parent(s)/legal guardian(s) agree that the subject will not participate in another interventional study while participating in the present study.
* Subject and subject's parent(s)/legal guardian(s) are willing and able to comply with the study requirements and with the concomitant medication restrictions.
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a female of childbearing potential
  * Female of child bearing potential who agrees to follow the contraceptive guidance from the time of informed consent/assent through at least 30 days after final IP administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final IP administration.
* Female subject must not donate ova starting at first dose of IP and throughout the study period and for 30 days after final IP administration.
* Male subject with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the treatment period and for 30 days after final IP administration.
* Male subject must agree not donate sperm during the treatment period and for 30 days after final IP administration.
* Male subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after final IP administration.

Additional Inclusion at Visit 3/Week 0 (Baseline)

* Subject must have a micturition frequency of at least 8 times (on average) per day, in the 7 days prior to visit 3/week 0 (baseline), as recorded in the bladder e-diary.
* Subject must have at least 1 daytime incontinence episode (on average) per day, during the 7-day period before visit 3/baseline, as recorded in the bladder e-diary.
* Subject whose symptoms are not satisfactorily controlled with urotherapy and still fulfills the inclusion/exclusion criteria will enter the study.

Exclusion Criteria:

Exclusion at Visit 1/Week -4 (Screening)

* Subject has extraordinary daytime only urinary frequency according to the ICCS definition.

  * This applies to a toilet-trained child who has the frequent need to void that is associated with small micturition volumes solely during the day.
  * The daytime voiding frequency is at least once per hour with an average voided volume of < 50% of expected bladder capacity (EBC) (typically 10% to 15%).
  * Incontinence is rare and nocturia is absent.
* Subject has an uroflow indicative of pathology other than OAB.
* Subject has monosymptomatic enuresis.
* Subject has dysfunctional voiding.
* Subject has bladder outlet obstruction, except if successfully treated.
* Subject has anatomical anomalies (surgically treated or untreated) that affect lower urinary tract function.
* Subject with hematuria on dipstick test. In the case of hematuria on dipstick test in a female during menstruation, the test can be repeated before randomization (after the end of menstruation).
* Subject with diabetes insipidus.
* Subject has kidney or bladder stones.
* Subject has suffered from chronic UTI or has had more than 3 UTIs in the 2 months prior to visit 1/week -4 (screening).
* Subject has stage 2 hypertension or subject has stage 1 hypertension that is not well controlled, as defined by the 2017 American Academy of Pediatrics Clinical Practice Guidelines.
* Subject has QT interval using Fridericia's correction formula (QTcF) > 440 msec on screening ECG, risk of QT prolongation (e.g., hypokalemia, long QT syndrome [LQTS] or family history of LQTS or exercise-induced syncope) or is currently taking medication known to prolong the QT interval.
* Subject's aspartate aminotransferase (AST) or alanine aminotransferase (ALT) is ≥ 2 × upper limit of normal (ULN) or total bilirubin (TBL) is ≥ 1.5 × ULN according to age and sex (subjects with Gilbert's syndrome are excepted from the bilirubin threshold).
* Subject has mild or moderate renal impairment (estimated glomerular filtration rate according to the modified Schwartz of < 60 mL/min per 1.73 m^2).
* Subject has a symptomatic (symptoms can include pain, fever, hematuria, new onset foul-smelling urine) UTI. Note: if the UTI is treated successfully (clinical recovery: confirmed by dipstick test and repeated dipstick test after 14 days [both should be negative]), the subject can be rescreened.
* Subject has a history or presence of any malignancy.
* Subject uses any drugs that are sensitive cytochrome P450 2D6 (CYP2D6) substrates with a narrow therapeutic index or sensitive P-glycoprotein (P-gp) substrates, or moderate or strong cytochrome CYP3A4/5 or P-gp inhibitors or inducers after the start of washout.
* Subject is using or has used prohibited prior and/or concomitant medication(s) that cannot be discontinued.
* Subject has known or suspected hypersensitivity to mirabegron or any components of the formulations used.
* Subject has participated in another clinical study (and/or subject has received any investigational therapy within 30 days (or 5 half-lives of the drug, or the limit set by national law, whichever is longer) prior to visit 1/week -4 (screening).
* Subject received urinary catheterization within 2 weeks prior to screening.
* Subject has constipation as defined by the Rome IV criteria that cannot be successfully treated prior to study entry.
* Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Subject has any condition that makes the subject unsuitable for study participation.

Additional Exclusion at Visit 3/Week 0 (Baseline)

* Subject has extraordinary daytime only urinary frequency according to the ICCS definition based on the bladder e-diary.
* Subject has monosymptomatic enuresis confirmed by the bladder e-diary.
* Subject has a maximum voided volume (morning volume excluded) > expected bladder capacity (EBC) for age ([age +1] × 30) in mL, based on the bladder e-diary.
* Subject has polyuria defined as voided urine volumes of > 40 mL/kg baseline body weight during 24 hours or > 2.8 L urine for a child weighing ≥ 70 kg (ICCS definition), based on bladder e-diary.
* Subject has PVR volume > 20 mL (lowest PVR volume result) as measured by ultrasonography.
* Subject suffers from a symptomatic (symptoms can include pain, fever, hematuria, new onset foul-smelling urine) urinary tract infection (UTI). Note: if a symptomatic UTI is present, all visit 3/week 0 (baseline) assessments must be postponed until the UTI is successfully treated (clinical recovery: confirmed by dipstick test and repeated dipstick test after 14 days [both should be negative]), and the urotherapy should continue. The postponed visit 3/week 0 (baseline) should be within 14 days of the intended visit 3/week 0 (baseline).
* Subject with hematuria on dipstick test. In the case of hematuria on dipstick test in a female during menstruation, the test can be repeated before randomization (after the end of menstruation).
* Subject has a pulse > 99th percentile for age.
* Subject has stage 2 hypertension or subject has stage 1 hypertension that is not well controlled, as defined by the 2017 American Academy of Pediatrics Clinical Practice Guidelines.
* Any reason that makes the subject unsuitable for study participation.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (15):
- Site BE32005, Ghent, Belgium
- Site FR33001, Marseille, France
- Site ML60002, Kuala Lumpur, Malaysia
- Site NO47001, Bergen, Norway
- Philippines (4):
  - Site PH63002, Angeles City
  - Site PH63004, Cebu City
  - Site PH63001, Quezon City
  - Site PH63005, Quezon City
- Russia (2):
  - Site RU70004, Moscow, Moscow
  - Site RU70001, Kazan', Tatarstan, Respublika
- South Korea (2):
  - Site KR82004, Yangsan, Gyeongsangnam-do
  - Site KR82001, Seoul, Seoul Teugbyeolsi
- Site TR90001, Bursa, Turkey (Türkiye)
- Site UA38007, Ivano-Frankivsk, Ukraine
- Site GB44004, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14573&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had received 4 weeks of urotherapy prior to randomization were enrolled in the study.
Pre-assignment Details: Standard urotherapy included information on and demystification of voiding function and dysfunction, instruction on voiding habits, lifestyle advice regarding fluid intake, prevention of constipation, recording of symptoms and voiding habits in bladder diaries and support via regular follow-up. Specific interventions included various forms of pelvic floor training, behavioral modification, electrical stimulation, catherization and biofeedback and elements of cognitive behavioral therapy.
Groups:
- Mirabegron (5 to < 12 Years): Participants aged 5 to < 12 years received initial dose of 25 mg of mirabegron orally once daily based on weight PED25 on day 1. Participants with a body weight ≥ 35 kg received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the PED50 based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
- Placebo (5 to < 12 Years): Participants aged 5 to < 12 years received placebo matched to mirabegron orally once daily based on weight PED25 on day 1. Participants with a body weight ≥ 35 kg received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the PED50 based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
- Mirabegron (12 to < 18 Years): Participants aged 12 to < 18 years received initial dose of 25 mg of mirabegron orally once daily based on weight PED25 on day 1. Participants with a body weight ≥ 35 kg received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the PED50 based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
- Placebo (12 to < 18 Years): Participants aged 12 to < 18 years received placebo matched to mirabegron orally once daily based on weight PED25 on day 1. Participants with a body weight ≥ 35 kg received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the PED50 based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
Period: Overall Study
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years) | Mirabegron (12 to < 18 Years) | Placebo (12 to < 18 Years)
Started | 11 | 12 | 2 | 1
Completed | 9 | 10 | 1 | 0
Not Completed | 2 | 2 | 1 | 1
Not completed — Protocol Violation | 1 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years) | Mirabegron (12 to < 18 Years) | Placebo (12 to < 18 Years) | Total
Number analyzed (Participants) | 11 | 12 | 2 | 1 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.4 (1.9) | 7.7 (1.7) | 16 (1.4) | 12 (NA) — Only 1 participant was analyzed, therefore, SD was not possible to calculate. | 8.8 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 2 | 0 | 11
  Male | 9 | 5 | 0 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 11 | 2 | 1 | 23
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 6 | 1 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 6 | 1 | 0 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Mean Number of Micturitions per 24 hour [Mean (Standard Deviation); unit: Micturitions per 24 hours] — A micturition was defined as any voluntary act of passing urine (excluding incontinence only episodes). The mean number of micturitions per 24 hours was calculated as the average number of times a participant urinated per day during the 7-day micturition diary period. Population: Participants in the SAF with available data were analyzed.
  Micturitions per 24 hours
    number analyzed (Participants) | 11 | 11 | 2 | 1 | 25
    (all) | 9.48 (4.53) | 9.72 (4.95) | 19.43 (3.16) | 9.29 | 10.37 (5.16)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12/EoT in Mean Number of Micturitions Per 24 Hours for Age Group 5 to <12 Years
Description: A micturition was defined as any voluntary act of passing urine (excluding incontinence only episodes). The mean number of micturitions per 24 hours was calculated as the average number of times a participant urinated per day during the 7-day micturition diary period. The analysis was performed with imputation of missing visit 7/week 12 data using the last observation carried forward (LOCF) method.
Time Frame: Baseline, week 12
Population: Full Analysis set: All participants who were randomized and received at least 1 dose of study drug and had at least 1 post baseline measurement for mean number of micturitions per 24 hours.
Measure: Least Squares Mean (Standard Error); unit: micturitions per 24 hours
Groups:
- Mirabegron (5 to < 12 Years): Participants aged 5 to < 12 years received initial dose of 25 milligram (mg) of mirabegron orally once daily based on weight (pediatric equivalent dose of 25 mg [PED25]) on day 1. Participants with a body weight ≥ 35 kilogram (kg) received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the pediatric equivalent dose of 50 mg [PED50] based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years)
Number analyzed (Participants) | 9 | 10
micturitions per 24 hours | -1.62 (0.89) | -3.84 (0.89)
Statistical Analysis 1: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); Analysis of Covariance (ANCOVA) was performed with change from baseline at week 12 Last Observation Carried Forward (LOCF) as response, treatment group, sex and geographical region as fixed effects and the mean number of micturitions per 24 hours at baseline as covariate; Test type: Superiority; p = 0.121, ANCOVA; LS Mean difference = 2.22, 90% CI 2-sided [-0.15 to 4.59], Standard Error of Mean 1.34

2. Secondary Outcome: Change From Baseline to Week 12/EoT in Mean Volume Voided Per 24 Hours for Age Group 5 to <12 Years
Description: Mean volume voided was derived from "Pee Volume" of the 2-day Weekend Episodic Diary. Mean volume voided per day was calculated as the sum of the volumes voided on that (valid diary) day divided by the number of times a volume was recorded on that day in the 2-day Weekend Episodic Diary. The analysis was performed with LOCF and without LOCF method.
Time Frame: Baseline, week 12
Population: Full Analysis Set with available data was analyzed.
Measure: Mean (Standard Deviation); unit: milliliter (mL)/24 hours
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years)
Number analyzed (Participants) | 8 | 8
milliliter (mL)/24 hours
  Week 12 (without LOCF) | 18.38 (33.67) | 24.55 (32.32)
  Week 12 (with LOCF) | 18.38 (33.67) | 24.55 (32.32)
Statistical Analysis 1: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); ANCOVA was performed with change from baseline at week 12 without LOCF as response, treatment group, sex and geographical region as fixed effects and the mean volume voided per 24 hours at baseline as covariate. Statistically significant treatment difference at 0.10 level for mirabegron vs placebo; Test type: Superiority; p = 0.430, ANCOVA; Mean Difference (Final Values) = -15.51, 90% CI 2-sided [-49.47 to 18.46], Standard Error of Mean 18.91
Statistical Analysis 2: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); ANCOVA was performed with change from baseline at week 12 with LOCF as response, treatment group, sex and geographical region as fixed effects and the mean volume voided per 24 hours at baseline as covariate. Statistically significant treatment difference at 0.10 level for mirabegron vs placebo; Test type: Superiority; p = 0.430, ANCOVA; Mean Difference (Final Values) = -15.51, 90% CI 2-sided [-49.47 to 18.46], Standard Error of Mean 18.91

3. Secondary Outcome: Change From Baseline to Week 12/EoT in Maximum Volume Voided (MVV) for Age Group 5 to <12 Years
Description: MVV data was derived from "Pee Volume" of the 2-day Weekend Episodic Diary. The MVV was the largest (non-zero) volume recorded over both of the 2 (valid) measuring days in the diary. The analysis was performed with LOCF and without LOCF method.
Time Frame: Baseline, week 12
Population: Full Analysis Set with available data was analyzed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years)
Number analyzed (Participants) | 8 | 8
mL
  Week 12 (without LOCF) | 26.00 (51.46) | 26.38 (60.75)
  Week 12 (With LOCF) | 26.00 (51.46) | 26.38 (60.75)
Statistical Analysis 1: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.935, ANCOVA; Mean Difference (Final Values) = 2.58, 90% CI 2-sided [-53.23 to 58.38], Standard Error of Mean 31.08
Statistical Analysis 2: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.935, ANCOVA; Mean Difference (Final Values) = 2.58, 90% CI 2-sided [-53.23 to 58.38], Standard Error of Mean 31.08

4. Secondary Outcome: Change From Baseline to Week 12/EoT in Mean Number of Daytime Incontinence Episodes Per 24 Hours for Age Group 5 to <12 Years
Description: A daytime incontinence episode was defined as the complaint of any involuntary leakage of urine during daytime hours. Daytime was defined as time between waking up in the morning and going to sleep later the same day or next day. The mean number of daytime incontinence episodes per 24 hours was calculated by taking the sum of all daytime urinary incontinence episodes recorded in the participant diary, divided by the number of valid diary days. The analysis was performed with LOCF and without LOCF method.
Time Frame: Baseline, week 12
Population: Full Analysis Set with available data was analyzed.
Measure: Mean (Standard Deviation); unit: incontinence episodes per 24 hours
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years)
Number analyzed (Participants) | 8 | 9
incontinence episodes per 24 hours
  Week 12 (without LOCF) | -1.29 (1.04) | -1.28 (1.73)
  Week 12 (with LOCF) | -1.20 (1.02) | -1.09 (1.74)
Statistical Analysis 1: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.073, ANCOVA; Mean Difference (Final Values) = -1.04, 90% CI 2-sided [-1.99 to -0.10], Standard Error of Mean 0.53
Statistical Analysis 2: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.044, ANCOVA; Mean Difference (Final Values) = -1.00, 90% CI 2-sided [-1.80 to -0.20], Standard Error of Mean 0.45

5. Secondary Outcome: Change From Baseline to Week 12/EoT in Mean Number of Nighttime Incontinence Episodes Per 24 Hours for Age Group 5 to <12 Years
Description: A nighttime incontinence episode was defined as the complaint of any involuntary leakage of urine during nighttime hours. Nightime was defined as time between between going to sleep on a day and waking up on the same or next day. The mean number of nighttime incontinence episodes per 24 hours was calculated by taking the sum of all nighttime urinary incontinence episodes recorded in the participant diary, divided by the number of valid diary days. The analysis was performed with LOCF and without LOCF method.
Time Frame: Baseline, week 12
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: incontinence episodes per 24 hours
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years)
Number analyzed (Participants) | 9 | 10
incontinence episodes per 24 hours
  Week 12 (without LOCF) | -0.64 (0.55) | -1.34 (1.51)
  Week 12 (with LOCF) | -0.64 (0.55) | -1.34 (1.51)
Statistical Analysis 1: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); ANCOVA as performed with change from baseline at week 12 without LOCF as response, treatment group, sex and geographical region as fixed effects and the mean number of daytime incontinence episodes per 24 hours at baseline as covariate. Statistically significant treatment difference at 0.10 level for mirabegron vs placebo; Test type: Superiority; p = 0.910, ANCOVA; Mean Difference (Final Values) = -0.05, 90% CI 2-sided [-0.74 to 0.64], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); ANCOVA as performed with change from baseline at week 12 with LOCF as response, treatment group, sex and geographical region as fixed effects and the mean number of daytime incontinence episodes per 24 hours at baseline as covariate. Statistically significant treatment difference at 0.10 level for mirabegron vs placebo; Test type: Superiority; p = 0.910, ANCOVA; Mean Difference (Final Values) = -0.05, 90% CI 2-sided [-0.74 to 0.64], Standard Error of Mean 0.39

6. Secondary Outcome: Change From Baseline to Week 12/EoT in Mean Number of Daytime Micturitions Per 24 Hours for Age Group 5 to <12 Years
Description: For a week day the daytime micturitions was derived from "Number of Times using the Toilet During the Day" was entered into the 5-day Week Diary. For a weekend day the daytime micturitions was derived from the number of times a "Pee in Toilet" or a "Pee in Toilet and Leakage" was entered into the 2-day Weekend Episodic Diary between the time the participant woke-up (exclusive). The total number of micturitions per weekend day was equal to the total number of times, in the diary, an amount of pee was recorded during daytime for that day. For each participant, the mean number of daytime micturitions was calculated as:
  Sum of the Number of Daytime Micturitions (per day) over the Valid Diary Days prior to Visit/Number of Valid Diary Days.
  The analysis was performed with LOCF and without LOCF method.
Time Frame: Baseline, week 12
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years)
Number analyzed (Participants) | 9 | 10
micturitions per 24 hours
  Week 12 (without LOCF) | -0.85 (2.67) | -3.21 (6.65)
  Week 12 (with LOCF) | -0.85 (2.67) | -3.21 (6.27)
Statistical Analysis 1: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); ANCOVA was performed with change from baseline at week 12 without LOCF as response, treatment group, sex and geographical region as fixed effects and the mean number of daytime micturitions per 24 hours at baseline as covariate. Statistically significant treatment difference at 0.10 level for mirabegron vs placebo; Test type: Superiority; p = 0.012, ANCOVA; Mean Difference (Final Values) = 2.48, 90% CI 2-sided [0.97 to 3.99], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); ANCOVA was performed with change from baseline at week 12 with LOCF as response, treatment group, sex and geographical region as fixed effects and the mean number of daytime micturitions per 24 hours at baseline as covariate. Statistically significant treatment difference at 0.10 level for mirabegron vs placebo; Test type: Superiority; p = 0.007, ANCOVA; Mean Difference (Final Values) = 2.46, 90% CI 2-sided [1.10 to 3.82], Standard Error of Mean 0.77

7. Secondary Outcome: Change From Baseline to Week 12/EoT in Number of Dry (Incontinence-free) Days Per 7 Days for Age Group 5 to <12 Years
Description: A dry (incontinence free) day was defined as a day where the response is "Dry" to the question "How was your Day" and to "How was your Night". For a weekend day a "Dry (incontinence free) Day" was defined a day where no "New pee or leakage" was reported. Let Ddry be the number of valid diary days where the response to both questions was "Dry". Let Dwet be the number of valid diary days where the response to one of the two questions or to both questions was "Wet". If (Ddry + Dwet) > 3, the number of dry days per 7 days was calculated as Ddry/(Ddry + Dwet)* 7, otherwise the value was missing.
  The analysis was performed with LOCF and without LOCF method.
Time Frame: Baseline, week 12
Population: Full Analysis Set with available data was analyzed.
Measure: Mean (Standard Deviation); unit: incontinence-free days
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years)
Number analyzed (Participants) | 9 | 9
incontinence-free days
  Week 12 (without LOCF): number analyzed (Participants) | 8 | 7
  Week 12 (without LOCF) | 3.12 (3.36) | 1.45 (2.33)
  Week 12 (with LOCF) | 2.94 (3.47) | 1.46 (2.18)
Statistical Analysis 1: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); Without LOCF: From a negative binomial regression model including treatment group, sex and region as factors and the log baseline rate of number of dry days (the log of the ratio of dry days at baseline and number of diary days at baseline) as covariate; Test type: Superiority; p = 0.105, Binomial regression; Rate ratio = 0.20, 90% CI 2-sided [0.04 to 1.02]
Statistical Analysis 2: Comparison: Mirabegron (5 to < 12 Years) vs Placebo (5 to < 12 Years); With LOCF: From a negative binomial regression model including treatment group, sex and region as factors and the log baseline rate of number of dry days (the log of the ratio of dry days at baseline and number of diary days at baseline) as covariate; Test type: Superiority; p = 0.111, Binomial regression; Rate ratio = 0.22, 90% CI 2-sided [0.05 to 1.05]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was any untoward medical occurrence in a participant administered a study drug and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug whether or not considered related to the study drug. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted a congenital anomaly/birth defect or other medically important event. A TEAE was defined as an AE observed after starting administration of the study drug until 30 days after last dose.
Time Frame: From first dose up to week 14
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years) | Mirabegron (12 to < 18 Years) | Placebo (12 to < 18 Years)
Number analyzed (Participants) | 11 | 12 | 2 | 1
Participants
  Treatment emergent adverse events | 5 | 7 | 1 | 1
  Serious treatment emergent adverse events | 0 | 0 | 1 | 1

9. Secondary Outcome: Change From Baseline in Post Void Residual (PVR) Volume
Description: PVR was assessed by ultrasonography.
Time Frame: Baseline, weeks 4, 12, 14
Population: SAF with available data was analyzed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years) | Mirabegron (12 to < 18 Years) | Placebo (12 to < 18 Years)
Number analyzed (Participants) | 10 | 10 | 2 | 1
mL
  Week 4: number analyzed (Participants) | 9 | 10 | 2 | 0
  Week 4 | -0.56 (11.59) | 8.80 (29.90) | -3.00 (9.90) |
  Week 12: number analyzed (Participants) | 8 | 7 | 1 | 1
  Week 12 | 1.63 (4.27) | 5.43 (12.79) | 5.00 (NA) — Only 1 participant was analyzed, therefore, SD was not possible to be calculated. | 0.00 (NA) — Only 1 participant was analyzed, therefore, SD was not possible to be calculated.
  Week 14 | 2.20 (8.44) | 11.0 (33.60) | 4.50 (0.71) | 0.00 (NA) — Only 1 participant was analyzed, therefore, SD was not possible to be calculated.

10. Secondary Outcome: Number of Participants With Study Drug Acceptability and Palatability for Tablets
Description: Participants evaluated the taste of the study drug/tablets by ticking 1 of the following categories: "Really Bad" (0), "Bad" (1), "Not Bad, Not Good" (2), "Good" (3) & "Really Good" (4). Participants evaluated the swallow of the study drug/tablets by ticking one of the following categories: "Really Difficult" (0), "Difficult" (1), "Not Difficult, Not Easy" (2), "Easy" (3) and "Really Easy" (4).
Time Frame: Week 12
Population: SAF with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years) | Mirabegron (12 to < 18 Years) | Placebo (12 to < 18 Years)
Number analyzed (Participants) | 3 | 1 | 2 | 0
Participants
  Taste: Really bad | 0 | 0 | 0 |
  Taste: Bad | 1 | 0 | 0 |
  Taste: Not Bad, Not Good | 1 | 1 | 2 |
  Taste: Good | 1 | 0 | 0 |
  Taste: Really Good | 0 | 0 | 0 |
  Swallow: Really Difficult | 0 | 0 | 0 |
  Swallow: Difficult | 0 | 0 | 0 |
  Swallow: Not Difficult, Not Easy | 0 | 0 | 1 |
  Swallow: Easy | 2 | 0 | 0 |
  Swallow: Really Easy | 1 | 1 | 1 |

11. Secondary Outcome: Number of Participants With Study Drug Acceptability and Palatability for Oral Suspension
Description: Participants evaluated the taste of the study drug/oral suspension by ticking 1 of the following categories: "Really Bad" (0), "Bad" (1), "Not Bad, Not Good" (2), "Good" (3) & "Really Good" (4). Participants evaluated the smell of the study drug/oral suspension by ticking 1 of the following categories: "Really Bad" (0), "Bad" (1),"Not Bad, Not Good" (2), "Good" (3) & "Really Good" (4). Participants evaluated the consumption of the study drug/oral suspension by ticking 1 of the following categories: "Really Difficult" (0),"Difficult" (1), "Not Difficult, Not Easy" (2), "Easy" (3) & "Really Easy" (4). Participants evaluated the preparation of the study drug/oral suspension by ticking 1 of the following categories: "Really Difficult" (0), "Difficult" (1), "Not Difficult, Not Easy" (2), "Easy" (3) & "Really Easy" (4).
Time Frame: Week 12
Population: SAF with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | Mirabegron (5 to < 12 Years) | Placebo (5 to < 12 Years) | Mirabegron (12 to < 18 Years) | Placebo (12 to < 18 Years)
Number analyzed (Participants) | 6 | 7 | 0 | 0
Participants
  Taste: Really Bad | 0 | 0 |  |
  Taste: Bad | 0 | 0 |  |
  Taste: Not Bad, Not Good | 4 | 6 |  |
  Taste: Good | 1 | 1 |  |
  Taste: Really Good | 1 | 0 |  |
  Smell: Really Bad | 0 | 0 |  |
  Smell: Bad | 0 | 0 |  |
  Smell: Not Bad, Not Good | 3 | 4 |  |
  Smell: Good | 0 | 2 |  |
  Smell: Really Good | 3 | 1 |  |
  Taking: Really Difficult | 0 | 0 |  |
  Taking: Difficult | 0 | 0 |  |
  Taking: Not Difficult, Not Easy | 0 | 1 |  |
  Taking: Easy | 4 | 5 |  |
  Taking: Really Easy | 2 | 1 |  |
  Preparing: Really Difficult | 0 | 0 |  |
  Preparing: Difficult | 0 | 0 |  |
  Preparing: Not Difficult, Not Easy | 0 | 2 |  |
  Preparing: Easy | 4 | 5 |  |
  Preparing: Really Easy | 2 | 0 |  |

12. Secondary Outcome: Pharmacokinetic (PK) of Mirabegron in Plasma: Maximum Concentration (Cmax)
Description: Maximum observed plasma concentration (Cmax).
Time Frame: Predose (1 hour prior) at weeks 4 and 12
Population: PK parameter calculation was not possible due to low number of samples collected.
Arm/Group | Mirabegron (5 to < 12 Years) | Mirabegron (12 to < 18 Years)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: PK of Mirabegron in Plasma: Time of the Maximum Concentration (Tmax)
Description: Time taken to reach Cmax (Tmax).
Time Frame: Predose (1 hour prior) at weeks 4 and 12
Population: PK parameter calculation was not possible due to low number of samples collected.
Arm/Group | Mirabegron (5 to < 12 Years) | Mirabegron (12 to < 18 Years)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: PK of Mirabegron in Plasma: Area Under Concentration-time Curve Over Dosing Interval (AUCtau)
Description: AUCtau is the measure of the plasma drug concentration from time zero to end of dosing interval. It is used to characterize drug absorption.
Time Frame: Predose (1 hour prior) at weeks 4 and 12
Population: PK parameter calculation was not possible due to low number of samples collected.
Arm/Group | Mirabegron (5 to < 12 Years) | Mirabegron (12 to < 18 Years)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: PK of Mirabegron in Plasma: Concentration Immediately Prior to Dosing (Ctrough)
Description: Trough level or trough concentration (Ctrough) in the concentration reached by the drug immediately before the next dose is administered.
Time Frame: Predose (1 hour prior) at weeks 4 and 12
Population: Pharmacokinetics Analysis Set included all participants who took at least 1 dose of study drug and contributed at least one pharmacokinetic sample in which the date and time of the sample and prior dose were known.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Mirabegron (12 to < 18 Years): Mirabegron (12 to < 18 years) Participants aged 12 to < 18 years received initial dose of 25 mg of mirabegron orally once daily based on weight PED25 on day 1. Participants with a body weight ≥ 35 kg received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the PED50 based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
Arm/Group | Mirabegron (5 to < 12 Years) | Mirabegron (12 to < 18 Years)
Number analyzed (Participants) | 8 | 1
ng/mL
  Week 4: number analyzed (Participants) | 7 | 1
  Week 4 | 3.18 (1.01) | 0.00 (NA) — Only 1 participant was analyzed, therefore, SD was not possible to be calculated.
  Week 12: number analyzed (Participants) | 8 | 0
  Week 12 | 12.68 (21.33) |

16. Secondary Outcome: PK of Mirabegron in Plasma: Apparent Total Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Predose (1 hour prior) at weeks 4 and 12
Population: PK parameter calculation was not possible due to low number of samples collected.
Arm/Group | Mirabegron (5 to < 12 Years) | Mirabegron (12 to < 18 Years)
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: PK of Mirabegron in Plasma: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F is influenced by the fraction absorbed.
Time Frame: Predose (1 hour prior) at weeks 4 and 12
Population: PK parameter calculation was not possible due to low number of samples collected.
Arm/Group | Mirabegron (5 to < 12 Years) | Mirabegron (12 to < 18 Years)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose up to week 14
Description: SAF
Groups:
- Mirabegron(5 to<12 Years): Participants aged 5 to < 12 years received initial dose of 25 mg of mirabegron orally once daily based on weight PED25 on day 1. Participants with a body weight ≥ 35 kg received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the PED50 based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
- Mirabegron(12 to<18 Years): Participants aged 12 to < 18 years received initial dose of 25 mg of mirabegron orally once daily based on weight PED25 on day 1. Participants with a body weight ≥ 35 kg received tablet and participants with a body weight< 35 kg or those who could not be dosed with the tablet received an oral suspension. At week 4, participants were up-titrated to the PED50 based on the given dose titration criteria up to week 12. Urotherapy continued throughout the study treatment period until week 12.
Arm/Group | Mirabegron(5 to<12 Years) | Placebo (5 to < 12 Years) | Mirabegron(12 to<18 Years) | Placebo (12 to < 18 Years)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 5/11 | 7/12 | 1/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron(5 to<12 Years) (N=11) | Placebo (5 to < 12 Years) (N=12) | Mirabegron(12 to<18 Years) (N=2) | Placebo (12 to < 18 Years) (N=1)
Diffuse axonal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron(5 to<12 Years) (N=11) | Placebo (5 to < 12 Years) (N=12) | Mirabegron(12 to<18 Years) (N=2) | Placebo (12 to < 18 Years) (N=1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT04641975/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT04641975/SAP_001.pdf